CLINICAL TRIAL: NCT00087997
Title: A Study of STA-4783 in Combination With Weekly Paclitaxel for Treatment of Patients With Soft Tissue Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4783-04
Record Dates: First submitted 2004-07-19; First posted 2004-07-23 (Estimated); Last update posted 2006-06-20 (Estimated); Status verified 2006-06

CONDITIONS: Soft Tissue Sarcoma
Keywords: sarcoma
MeSH Terms: conditions — Sarcoma | interventions — elesclomol

INTERVENTIONS:
Drug: STA-4783

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of an experimental study drug (STA-4783) combined with an approved cancer medicine, paclitaxel, in the treatment of soft tissue sarcomas. Paclitaxel (Taxol®) has been approved and used in the United States since 1992.

DETAILED DESCRIPTION:
STA-4783 is a taxane potentiator, enhancing the effect of antitumor response of paclitaxel. In an attempt to improve efficacy, paclitaxel is sometimes used in combination with other anticancer agents. When paclitaxel is combined with other anticancer agents, although response rate is usually increased, side effects are usually increased as well. There is an urgent need for agents that can enhance the antitumor effects of paclitaxel without further increasing undesirable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older with histologic diagnosis of soft tissue sarcoma
* Must have disease not suitable for curative resection
* Must have failed >1 first line treatment with evidence of progression. Adjuvant therapy does not count as 1st line therapy unless recurrence occurs within 6 months of administration
* Must have ability to understand and the willingness to sign a written informed consent document
* Must have Eastern Cooperative Oncology Group (ECOG) performance status of < 2
* Must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* At least 4 weeks have passed since the last chemotherapy, immunotherapy, or radiation therapy
* There must be measurable disease outside the radiotherapy fields or progression of the indicator lesions within the field since the completion of the radiotherapy
* Must have a life expectancy of greater than 12 weeks
* Must have clinical laboratory values at screening as defined below:
* Hemoglobin >9 g/dL,
* Absolute neutrophil count >1500/mm3,
* Platelet count >100,000/mm3,
* Creatinine <1.5 X ULN,
* Bilirubin <1.5 X ULN,
* Asparate aminotransferase and alanine aminotransferase <2.5 X ULN (<5 X ULN in presence of liver metastases)

Exclusion Criteria:

* Female patients who are pregnant or breast feeding
* Patients of childbearing potential not using or not willing to use a barrier method of contraception
* Prior malignancy other than soft tissue sarcoma (STS) within the last 5 yrs with the exception of:

  * Adequately treated in situ carcinoma of the cervix uteri;
  * Basal or squamous cell carcinoma of the skin
* Presence of a clinically significant and uncontrolled infection
* Presence of >Grade 2 neuropathy
* Symptomatic central nervous system metastases within last 8 weeks or on corticosteroids for CNS symptom management
* Presence of clinically significant arrythmias
* Presence of a serious concurrent illness or other conditions (e.g., psychological, family, sociological, or geographical circumstances) that do not permit adequate follow-up and compliance with the protocol
* History of severe hypersensitivity reactions to taxanes or cremaphore in spite of premedication
* Use of any investigational agents within 4 weeks prior to the first dose of study drug(s)
* Major surgery within 2 weeks of screening
* Radiation treatment in past >25% of bone marrow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-07; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (27):
- United States (26):
  - Arizona Cancer Center, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - UCLA, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Department of Medicine, Chicago, Illinois
  - Via Christi Regional Med. Center (Wichita CCOP), Wichita, Kansas
  - University of Louisville Hospital, Louisville, Kentucky
  - Feist-Weiller Cancer Center, Shreveport, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYU Cancer Institute Clinical Center, New York, New York
  - Herbert Irving Cancer Center, New York, New York
  - Carolinas Medical Center/Blumenthal Cancer Center, Charlotte, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The West Clinic, Memphis, Tennessee
  - The Sarah Cannon Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Mount Sinai Hospital, Toronto, Ontario, Canada